CLINICAL TRIAL: NCT00051532
Title: Seocalcitol Versus Placebo in Advanced Hepatocellular Carcinoma. Efficacy of Seocalcitol (EB 1089) Enteric-Coated Capsules (5ug) or Placebo in the Treatment of Patients With Hepatocellular Carcinoma Not Amenable to Curative Treatment
Brief Title: Seocalcitol Versus Placebo in Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Masking: Double | Purpose: Other
Other Study IDs: EBC 9801 INT; EBC 9801 INT
Record Dates: First submitted 2003-01-13; First posted 2003-01-14 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2005-04

CONDITIONS: Liver Neoplasms
Keywords: hepatocellular; carcinoma; liver; cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma; Neoplasms | interventions — seocalcitol

INTERVENTIONS:
Drug: Seocalcitol

SUMMARY:
The purpose of the study is to determine whether seocalcitol is effective in the treatment of advanced primary liver cancer (hepatocellular carcinoma [HCC]).

ELIGIBILITY:
Inclusion Criteria:

* Hospital in- or out-patients
* Either sex
* Aged 18-75 years
* With hepatocellular carcinoma, verified by histology/cytology, which is not amenable to curative treatment or transplantation.
* Patients must have measurable disease, and be classifiable as to Barcelona Clinic Liver Cancer (BCLC) stage 0, as described in Llovet JM et al. Hepatology 1999;29:62-67.

Exclusion Criteria:

* Patients treated with chemotherapy or other anti-cancer therapy within 4 weeks before visit 1
* Patients with another primary tumor, except for basocellular carcinoma of the skin or in situ carcinoma of the cervix, within the last 2 years
* A history of renal stone(s)
* A life expectancy of < 3 months
* World Health Organization (WHO) performance status 3 or 4
* Okuda stage III.
* Patients with hypercalcemia, or other clinically important laboratory abnormalities
* Patients with previous/current calcium metabolic disease, taking calcium-lowering therapy, or medication known to affect systemic calcium metabolism are also excluded.
* All patients must give their signed informed consent to join the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 1999-09; Study Completion 2004-05

PRIMARY OUTCOMES:
Overall survival, defined as the time from start of treatment to death

SECONDARY OUTCOMES:
HCC-specific survival from start of treatment
Time to response from start of treatment (complete or partial response)
Proportion of patients who achieve partial/complete response
Time to progression measured from start of treatment
Duration of complete response in patients showing a complete response, measured from the first date when absence of disease was recorded until the first date of disease progression was recorded
Duration of partial response in patients showing partial response, measured from first date when partial response was recorded until the first date at which disease progression was observed
Duration of stable disease measured from start of treatment until the first date where either progression or partial/complete response was observed
Change(s) in tumour size
Change in tumour marker
Number of days of hospitalisation (in-patient care)
Quality of life
Adverse events
Change in laboratory values
Dose of seocalcitol (seocalcitol treated patients)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Hvidberg, MSc Pharm, PhD, Study Director — LEO Pharma
Locations (5):
- E.g. University Health Network Toronto General Hospital (numerous facilities are recruiting in Canada), Toronto, Alberta, Canada
- E.g. Notre-Dame de Bon Secours, Service d´Hepato-Gastro-Enterologie (numerous facilities are recruiting in France), Metz, France
- E.g. Osp. Maggiore, Policlinico di Milano (numerous facilities are recruiting in Italy), Milan, Italy
- E.g. Hospital Clinic Provincial de Barcelona (numerous facilities are recruiting in Spain), Barcelona, Spain
- E.g. The University of Edinburgh Royal Infirmary (numerous facilities are recruiting in UK), Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en